CLINICAL TRIAL: NCT01829204
Title: A Prospective Longitudinal Data Bank Creation to Study Vaginal Conditions With a Novel Diagnostic Approach
Brief Title: Prospective Data Bank Creation to Study Vaginal Conditions
Acronym: CRIPB-13-002
Status: Recruiting | Type: Observational
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Other Study IDs: L13-054
Record Dates: First submitted 2013-04-08; First posted 2013-04-11 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Vulvodynia; Mycoses; Bacterial Vaginosis; Preterm Labor
MeSH Terms: conditions — Vulvodynia; Mycoses; Vaginosis, Bacterial; Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Non pregnant asymptomatic: Asymptomatic, non-pregnant, healthy women ages 21 to 75 years with no previous history of any chronic or recurrent vulvovaginal condition who attend our clinical offices for their annual well-woman physical examination
- Non pregnant symptomatic: Non-pregnant women ages 12 to 75 years being evaluated for any gynecological vulvovaginal condition.
- Pregnant asymptomatic: Pregnant women ages 12 to 75 years who are both asymptomatic and healthy
- Pregnant symptomatic: Pregnant women ages 12 to 75 who have any gynecological vulvovaginal condition

SUMMARY:
The purpose of this study is to identify and elucidate the pattern and perhaps role of atypical proteins, cytokines and vaginal microbial flora in the pathogenic mechanisms involved in the development of vulvodynia, recurrent fungal and bacterial vaginosis and preterm labor.

DETAILED DESCRIPTION:
Our approach specifically targets the evaluation of the proteins and cytokines present and the bacteriological analysis of the microflora in the vaginal milieu.

Conjectures:

* An initial insult in the vagina (possibly involving a bacterial, viral or fungal organism or their products) causes modifications in the vaginal milieu
* The vaginal milieu responds to the insult by developing an inflammatory reaction characterized by cytokine and protein production
* Long lasting or repetitive insults maintain biochemical changes in the vaginal milieu producing a reaction, chemical irritation or micro flora alteration by changes in proteins and/or abnormal protein production
* Those changes eventually result in hypersensitivity, irritation, burning, and pain manifested in patients with vulvodynia. And those changes may also result in the recurrence of fungal or bacterial infections
* Those changes may also contribute to initiate the cascade of premature events conducting to cervical effacement and dilation observed in preterm labor

The conjectures will be investigated by using a multidisciplinary approach including: microbiology, proteomics and cytokines evaluation of the vaginal milieu. Specifically we will be comparing an asymptomatic female population to serve as a baseline to patients affected by vulvodynia, recurrent fungal or bacterial vaginosis and/or pregnancy.

This is a prospective, descriptive study of about 550 women age 12 to 75 years. There will be four groups: 1) Asymptomatic healthy women, 2) Women being seen for any gynecological vulvovaginal condition, and 3) Pregnant women who are asymptomatic and healthy, and 4) Pregnant women have any gynecological vulvovaginal condition.

We will evaluate the following:

* Types of cytokines normally present in women and in patients with vulvodynia, recurrent fungal and bacterial vaginosis and preterm labor
* Normal microbiology flora in women and variations present in the vaginal milieu in these patients
* The presence of normal and atypical proteins in the vaginal milieu of healthy women and patients with vulvodynia, recurrent fungal and bacterial vaginosis and preterm labor
* Informed consent will be obtained and documented for participation in the study
* Comprehensive history assessment of environmental factors, topical vulvovaginal issues and co morbid conditions as defined in the exclusion criteria.
* Pelvic examination to obtain two samples via cotton swabs for proteomics, cytokines, vaginal lactobacillus from vaginal secretions.

A. Swab procedure:

The cotton swabs (2) will be introduced only in the middle vagina, one at the time, no other areas will be sampled.

B. Swab processing One swab will be placed in a special room temperature solution. This de-identified swab will be mailed for Lactobacillus.

The second de-identified swab is to be place in 2 separated micro-containers in Liquid Nitrogen Containers (one for cytokines and one for Proteomics). When 50 samples are completed they will be processed at TTUHSC Permian Basin campus, with the Proteomics testing being done in Lubbock.

Therefore, there are 3 samples, each processed differently. Data will be recorded in a confidential manner with no personal identifiers, only an assigned study subject number. As such, the de-identified data may serve as a database for additional studies. The computer used will belong to TTUHSC and be password protected, access limited to only authorized personnel. Consent forms will be stored separately from the study data in the research office.

ELIGIBILITY:
Inclusion Criteria:

* All patients willing to participate, and give informed consent, and
* Asymptomatic, non-pregnant, healthy women ages 21 to 75 years with no previous history of any chronic or recurrent vulvovaginal condition who attend our clinical offices for their annual well-woman physical examination.
* Non-pregnant women ages 21 to 75 years being evaluated for any gynecological vulvovaginal condition.
* Pregnant women ages 21 to 75 years who are both asymptomatic and healthy
* Pregnant women ages 21 to 75 who have any gynecological vulvovaginal condition

Exclusion Criteria:

* Asymptomatic patients ages < 21 or > 75, or symptomatic patients ages < 21 or > 75 years.
* Patients diagnosed with cancer or having any medical condition that is not under control including: diabetes mellitus, hypertension, collagen disease, hemoglobinopathy, renal insufficiency, depression, anxiety, psychosis and panic attacks
* Patients unable to follow the protocol or unwilling to participate

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients willing to participate, and give informed consent, and Asymptomatic, non-pregnant, healthy women ages 21 to 75 years with no previous history of any chronic or recurrent vulvovaginal condition who attend our clinical offices for their annual well-woman physical examination.
  2-Non-pregnant women ages 21 to 75 years being evaluated for any gynecological vulvovaginal condition.
  Pregnant women ages 21 to 75 years who are both asymptomatic and healthy Pregnant women ages 21 to 75 who have any gynecological vulvovaginal condition
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2013-04; Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Cytokines Determination | one time for all except pregnant patients 4 times 12 months
  To determine types of cytokines normally present in women's vagina and in patients with vulvodynia, recurrent fungal and bacterial vaginosis and preterm labor

SECONDARY OUTCOMES:
Proteins Determination | one time for all except pregnant patients 4 times 12 months
  The vaginal milieu will respond to the insult by developing an inflammatory reaction characterized by protein production (in terms of increased protein concentration according to the Bradford protein assay).
Lactobacillus determination | one time for all except pregnant patients 4 times 12 months
  Long lasting or repetitive insults maintain biochemical changes in the vaginal milieu producing lactobacillus microflora alteration.

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Galloway, DO, Principal Investigator — TTUHSC PB
Locations (1):
- TTUHSC Permian Basin, Midland, Texas, United States

REFERENCES:
- [Background] Verstraelen H, Verhelst R, Claeys G, De Backer E, Temmerman M, Vaneechoutte M. Longitudinal analysis of the vaginal microflora in pregnancy suggests that L. crispatus promotes the stability of the normal vaginal microflora and that L. gasseri and/or L. iners are more conducive to the occurrence of abnormal vaginal microflora. BMC Microbiol. 2009 Jun 2;9:116. doi: 10.1186/1471-2180-9-116. PMID 19490622
- [Background] Ventolini G, Barhan SM. Vulvodynia. Dermatol Online J. 2008 Jan 15;14(1):2. PMID 18319019
- [Background] Ventolini G, Barhan S, Duke J. Vulvodynia, a step-wise therapeutic prospective cohort study. J Obstet Gynaecol. 2009 Oct;29(7):648-50. doi: 10.1080/01443610903095882. PMID 19757274
- [Background] Ventolini G. Measuring treatment outcomes in women with vulvodynia. J Clin Med Res. 2011 Apr 4;3(2):59-64. doi: 10.4021/jocmr526w. PMID 21811531
- [Background] Ventolini G. Vulvar pain: Anatomic and recent pathophysiologic considerations. Clin Anat. 2013 Jan;26(1):130-3. doi: 10.1002/ca.22160. Epub 2012 Sep 5. PMID 22951941
- [Background] Omoigui S. The biochemical origin of pain: the origin of all pain is inflammation and the inflammatory response. Part 2 of 3 - inflammatory profile of pain syndromes. Med Hypotheses. 2007;69(6):1169-78. doi: 10.1016/j.mehy.2007.06.033. Epub 2007 Aug 28. PMID 17728071
- [Background] Traisnel G, Lablanche JM, Fourrier JL, Marquand A, Bertrand ME. [Reproducibility of the exercise test and coronary vasomotor tonus]. Arch Mal Coeur Vaiss. 1988 Jun;81(6):765-72. French. PMID 3144947
- See also: Clinical Research Institute TTUHSC — http://www.ttuhsc.edu/clinicalresearch/